CLINICAL TRIAL: NCT06749847
Title: HPV Self-sampling in the General Population: Efficacy, Feasibility, Acceptability and Cost-effectiveness
Brief Title: HPV Self-sampling in the General Population
Acronym: MIRABELLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Centre Régional de Coordination des Dépistages des Cancers de Grand Est (Unknown); Central Hospital, Nancy, France (Other); CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IEC/24-01; 2023-215 (Other Grant/Funding Number: INCa)
Record Dates: First submitted 2024-12-13; First posted 2024-12-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; screening program; pilot project; randomised control trial; France
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a three-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Outreach (Experimental): Women receive invitation letter with HPV self-sampling kit; Direct mailing of HPV self-sampling kit; Women receive HPV self-sampling kit with instructions; SMS reminder at 3 months if no participation; Assistance provided for triage cytology if HPV positive.
  Interventions: Other: Women receive invitation letter with HPV self-sampling kit
- Choice (Experimental): Women receive an invitation letter offering a choice between ordering a free self-sampling kit or visiting a healthcare provider.
  Option between self-sampling and healthcare provider: women can choose testing method. If self-sampling chosen, kit sent to home. SMS reminder at 3 months if no participation.
  Interventions: Other: Women receive invitation letter with choice of ordering a free self-sampling kit or visit healthcare provider
- Control arm (No Intervention): Standard invitation to visit healthcare provider for cervical cancer screening. Standard screening procedure. Follow standard organized screening program procedure. HPV self-sampling offered at 12-month reminder if no participation.

INTERVENTIONS:
Other: Women receive invitation letter with HPV self-sampling kit — Direct mailing of HPV self-sampling kit. Women receive HPV self-sampling kit with instructions. SMS reminder at 3 months if no participation. Assistance provided for triage cytology if HPV positive.
  Arms: Outreach
Other: Women receive invitation letter with choice of ordering a free self-sampling kit or visit healthcare provider — Option between self-sampling and healthcare provider: women can choose testing method. If self-sampling chosen, kit sent to home. SMS reminder at 3 months if no participation.
  Arms: Choice

SUMMARY:
A randomized controlled trial comparing three strategies for cervical cancer screening: direct mailing of HPV self-sampling kit ("Outreach" arm), choice between self-sampling or healthcare provider sampling ("Choice" arm), and standard care (control arm) in two French departments.

DETAILED DESCRIPTION:
In France, over 3,000 women are diagnosed annually with cervical cancer and 1,100 die from it, despite organized screening programs. The national screening coverage rate of 59% (2018- 2020) remains well below the European Union's recommended target of 70% and even further from the French Cancer Plan 2014-2019 objective of 80%. This study evaluates two innovative strategies to improve participation rates in two French departments (Marne and Aube). Eligible women aged 30-65 years will be randomized into three arms. The "Outreach" arm receives HPV self-sampling kit directly at home with SMS reminder at 3 months if no participation. The "Choice" arm can choose between ordering a self-sampling kit or visiting a healthcare provider with SMS reminder at 3 months if no participation. The control arm follows standard procedure with self-sampling offered at 12-month reminder. Women with positive HPV self-sampling tests will be followed for triage cytology, with assistance provided for appointments in the "Outreach" arm and reminders at 6 months post-positive result in the "Choice" arm. The study assesses participation rates, triage completion rates, feasibility, acceptability, and cost-effectiveness of these strategies. If successful, findings could inform modifications to the national organized screening program.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 to 65 years old
* Living in the study area (Departments of Marne and Aube, France)
* At moderate risk of cervical cancer, i.e. eligible to the organised programme and receiving the first invitation of the screening round (not a reminder letter)

Exclusion Criteria:

* Outside the target age (less than 30 years old, or 66 years old and more)
* Already participating in the current screening round
* Total hysterectomy
* History of cervical cancer
* Current follow-up for abnormal cervical screening result or cervical lesions

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6000 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Participation rate in cervical cancer screening | 18 months after invitation

SECONDARY OUTCOMES:
Triage cytology completion rate after positive HPV test | 6 months after positive result
HPV positivity rate | 12 months after invitation
Invalid result rate | 18 months
Time from HPV-positive result to completion of cytological triage | 18 months
Women's acceptability of HPV self-sampling | 24 months
  Qualitative assessment through semi-structured interviews with 40 women to assess women's acceptability of HPV self-sampling
Cost-effectiveness of screening strategies | 24 months
  Costs will be estimated using an ingredients approach whereby resources used for the respective interventions (' Outreach ' and ' Choice' strategies) are identified and valued. The analysis will include all costs incurred by the screening program, including invitation materials, self-sampling kits, laboratory testing, result communication, and follow-up coordination. The incremental cost-effectiveness ratios (ICERs) will be calculated as the mean difference in total costs between each intervention arm and the control arm, divided by the mean difference in screening participation rates. Results will be expressed in euros per percentage change in screening participation.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie BERTRAND-BRICE, MD, Principal Investigator — Regional Cancer Screening Coordinating Centre, Marne site; Christine CLAVEL CRAVOISIER, Professor, Principal Investigator — CHU REIMS; Hamza ACHIT, PhD, Principal Investigator — CHRU Nancy; Farida SELMOUNI, PhD, Principal Investigator — International Agency for Research on Cancer; Catherine SAUVAGET, MD, PhD, Principal Investigator — International Agency for Research on Cancer
Locations (2):
- France (2):
  - Regional Cancer Screening Coordinating Centre, Aube site, Troyes, Aube
  - Regional Cancer Screening Coordinating Centre, Marne site, Reims, Marne

IPD SHARING:
Plan to Share IPD: No